CLINICAL TRIAL: NCT04773990
Title: Efficacy of Balance Training by Biodex Balance System on Gait Parameters and Balance in Patients With RLAS
Brief Title: Efficacy of Balance Training by BBS on Gait Parameters and Balance in Patients With RLAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Collaborators: Cairo University (Other)
Responsible Party: Principal Investigator, Hadeer Gamal Abd-Elmaboud Maghraby, Demonstrator at Department of musculoskeletal disorders and it's surgeries, MTI University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: RLAS
Record Dates: First submitted 2021-02-11; First posted 2021-02-26 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Ankle Sprains
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Fifty subjects (power analysis) of both gender diagnosed with recurrent lateral ankle sprain patients will be assigned randomly into 2 groups.
  * Group (A) will receive biodex balance training
  * Group (B)will receive a physical therapy exercise protocol only
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Other): Group (A) twenty-five patients will receive biodex balance training
  Interventions: Device: Biodex Balance System; Other: specific physical therapy exercise program
- Controlled Group (Other): twenty-five patients will receive a physical therapy exercise protocol
  Interventions: Other: specific physical therapy exercise program

INTERVENTIONS:
Device: Biodex Balance System — Subjects will receive several unique training modules using biodex
  Other Names: BBS
  Arms: Experimental Group
Other: specific physical therapy exercise program — Subjects will receive recommended PT program

SUMMARY:
This study will be conducted to find out the effect of adding balance training on gait parameters, balance, and Sensory Interaction

DETAILED DESCRIPTION:
LAS are not benign injuries. As many as 4 in 10 individuals will develop chronic ankle instability (CAI) after a first-time sprain, More than half of patients with osteoarthritis (OA) of the ankle report a history of a sport-related ankle injury, and 85% of those are LAS.

ELIGIBILITY:
Inclusion Criteria:

* The patient will be referred to the outpatient clinic of the orthopedic department, Faculty of physical therapy, MTI University. with a confirmed diagnosis of recurrent Lateral ankle sprain grade II
* Subjects will be excluded if they had one of the following criteria:

Previous musculoskeletal injury to the lower limb or lumbar spine including a fracture, a sprain, or an unstable joint other than the injured ankle.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — 25 male , 25 female
Enrollment: 50 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Cadence | Before Treatment and after 6 weeks of treatment
  Change in Cadence measurements using Walkway Gait System.
Gait time | Before Treatment and after 6 weeks of treatment
  Change in Gait time measurements using Walkway Gait System.
Clinical Test of Sensory Integration | Before Treatment and after 6 weeks of treatment
  Change in Clinical Sensory Integration test measurements using Biodex balance System.

CONTACTS AND LOCATIONS:
Locations (1):
- Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No